CLINICAL TRIAL: NCT04999540
Title: Trial of Tucidinostat in Combination With Fulvestrant in Patients With Hormone-receptor Positive Advanced Breast Cancer
Brief Title: Tucidinostat and Fulvestrant in Hormone-receptor Positive Advanced Breast Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Guangdong Women and Children Hospital (Other)
Responsible Party: Principal Investigator, Anqin Zhang, Chief Physician, Guangdong Women and Children Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GDWCH-001
Record Dates: First submitted 2021-07-31; First posted 2021-08-11 (Actual); Last update posted 2021-08-11 (Actual); Status verified 2021-08

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — N-(2-amino-5-fluorobenzyl)-4-(N-(pyridine-3-acrylyl)aminomethyl)benzamide; Fulvestrant

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tucidinostat + Fulvestrant (Experimental): Patients receive 30 mg Chidamide twice per week. Fulvestrant 500mg (2 syringes of Fulvestrant 250mg), Fulvestrant 500 mg i.m. every 28 (+/- 3) days plus an additional 500 mg on day 14 (+/-3) of first month only.
  Courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Tucidinostat; Drug: Fulvestrant

INTERVENTIONS:
Drug: Tucidinostat — 30 mg, administered orally twice per week (BIW)
Drug: Fulvestrant — Fulvestrant was supplied as a castor oil based solution in clear neutral glass pre-filled syringes. Each syringe will contain 250 mg of fulvestrant in 5 ml.

SUMMARY:
The purpose of the study is evaluate the efficacy and safety of tucidinostat in combination with fulvestrant in patients with hormone-receptor positive advanced breast cancer.

DETAILED DESCRIPTION:
Hormone-receptor positive breast cancer is the most common subtype in breast cancer. Tucidinostat is an oral subtype-selective histone deacetylase inhibitor, which showed preliminary signs of encouraging anti-tumour activity in patients with advanced hormone-receptor positive breast cancer in the previous studies. The aim of this study is to evaluate the efficacy and safety of Tucidinostat in combination with fulvestrant in patients with recurrent or metastatic hormone-receptor positive breast cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Female patients aged 18-75 years (including cutoff value);
2. The disease condition is inoperable, recurrent breast cancer, or metastatic breast cancer;
3. Histological or cytological confirmation of hormone receptor-positive [estrogen receptor (ER) positive and progesterone receptors (PgR) positive or negative] breast cancer;
4. At least one measurable lesion according to RECIST 1.1;
5. Prior treatment: have not received systemic chemotherapy for recurrent or metastatic breast cancer;
6. Eastern Cooperative Oncology Group Performance Status of 0-1;
7. Adequate function of major organs meets the following requirements):

   Absolute Neutrophils count≥ 1.5×10^9/L; Platelets count≥ 90×10^9/L; Hemoglobin ≥ 90g/L; Total bilirubin≤ 1.5 × the upper limit of normal (ULN); ALT and AST ≤ 2.5 × ULN; BUN and Cr ≤ 1.5 × ULN; Left ventricular ejection fraction (LVEF) ≥ 50%; QTcF(Fridericia correction) ≤ 470 ms; International normalized ratio(INR)≤1.5 × ULN; activated partial thromboplastin time(APTT) ≤ 1.5 × ULN;
8. Life expectancy ≥ 3 months;
9. Have signed informed consent.

Exclusion Criteria:

1. Patients have untreated central nervous system (CNS) metastases;
2. Patients with no measurable lesion according to RECIST 1.1;
3. Patients with bilateral breast cancer;
4. Patients with human epidermal growth factor receptor-2 (Her-2) positive;
5. Recurrent or metastatic disease occurs within 2 years during adjuvant endocrine therapy;
6. Patients previously received systemic chemotherapy for recurrent or metastatic breast cancer;
7. Patients previously received any HDAC inhibitor or fulvestrant treatment;
8. There are ascites, pleural effusion, pericardial effusion with clinical symptoms at baseline, those who need drainage, or those who have undergone drainage of serous effusion within 4 weeks before the first dose;
9. Inability to swallow, intestinal obstruction or other factors affecting the administration and absorption of the drug;
10. Patients with other invasive malignancies within 5 years or at the same time, with the exception of curatively-treated basal cell or squamous cell carcinoma of the skin or cervical carcinoma in situ;
11. Patients with a history of allergies to the drug components of this regimen;
12. Patients with active HBV and HCV infection; stable hepatitis B after drug treatment (HBV virus copy number is higher than the upper limit of reference value) and cured hepatitis C patients (HCV virus copy number exceeds the lower limit of detection method) can be included;
13. Patients with a history of immunodeficiency, including HIV positive, or other acquired or congenital immunodeficiency disease, history of organ transplantation;
14. Patients have uncontrolled or significant cardiovascular disease, including: Myocardial infarction (< the last 12 months); Uncontrolled angina (< the last 6 months); Congestive heart failure (< the last 6 months), or Left Ventricular Ejection Fraction (LVEF) < 50% prior to study entry;
15. Any mental or cognitive disorder, that would interfere the ability to understand the informed consent document or the operation and compliance of study;
16. Any other condition which is inappropriate for the study in the opinion of the investigators.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Estimated)
Dates: Start 2021-11-01 (Estimated); Primary Completion 2023-12-01 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | From date of treatment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 3 years.
  PFS was defined as the time from treatment until objective disease progression according to Response Evaluation Criteria in Solid Tumours version 1.1 (RECIST 1.1), or death by any cause, whichever is first met.

SECONDARY OUTCOMES:
overall survival (OS) | Time from treatment to death from any cause, assessed up to 3 years.
  Defined as from the date of treatment to date of death, irrespective of cause.
Objectivel response rate (ORR) | Response is assessed once every 8 weeks, from the day of treatment to the date of first documented progression, assessed up to 3 years.
  Defined as numbers of patients achieved complete response and partial response of treatment.
Duration of response (DOR) | From the day of treatment to the date of first documented progression, assessed up to 3 years.
  Defined as from the first date when criteria for response is met until the first date when the criteria for progression or death is met.
4.Clinical Benefit Rate (CBR) | From the day of treatment to the date of first documented progression, assessed up to 3 years.
  ORR is defined as percentage of participants with Complete Response, Partial Response or Stable Disease≥24 weeks, assessed by the investigators according to the RECIST v1.1.
Adverse event(AE) | From the day of treatment to the date of first documented progression, assessed up to 3 years.
  Adverse event related to treatment.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Osborne CK, Schiff R. Mechanisms of endocrine resistance in breast cancer. Annu Rev Med. 2011;62:233-47. doi: 10.1146/annurev-med-070909-182917. PMID 20887199
- [Background] Saxena NK, Sharma D. Epigenetic Reactivation of Estrogen Receptor: Promising Tools for Restoring Response to Endocrine Therapy. Mol Cell Pharmacol. 2010;2(5):191-202. PMID 21499573
- [Background] Turner NC, Ro J, Andre F, Loi S, Verma S, Iwata H, Harbeck N, Loibl S, Huang Bartlett C, Zhang K, Giorgetti C, Randolph S, Koehler M, Cristofanilli M; PALOMA3 Study Group. Palbociclib in Hormone-Receptor-Positive Advanced Breast Cancer. N Engl J Med. 2015 Jul 16;373(3):209-19. doi: 10.1056/NEJMoa1505270. Epub 2015 Jun 1. PMID 26030518
- [Background] Goetz MP, Toi M, Campone M, Sohn J, Paluch-Shimon S, Huober J, Park IH, Tredan O, Chen SC, Manso L, Freedman OC, Garnica Jaliffe G, Forrester T, Frenzel M, Barriga S, Smith IC, Bourayou N, Di Leo A. MONARCH 3: Abemaciclib As Initial Therapy for Advanced Breast Cancer. J Clin Oncol. 2017 Nov 10;35(32):3638-3646. doi: 10.1200/JCO.2017.75.6155. Epub 2017 Oct 2. PMID 28968163
- [Background] Falkenberg KJ, Johnstone RW. Histone deacetylases and their inhibitors in cancer, neurological diseases and immune disorders. Nat Rev Drug Discov. 2014 Sep;13(9):673-91. doi: 10.1038/nrd4360. Epub 2014 Aug 18. PMID 25131830
- [Background] Jones PA, Issa JP, Baylin S. Targeting the cancer epigenome for therapy. Nat Rev Genet. 2016 Sep 15;17(10):630-41. doi: 10.1038/nrg.2016.93. PMID 27629931
- [Background] Shi Y, Dong M, Hong X, Zhang W, Feng J, Zhu J, Yu L, Ke X, Huang H, Shen Z, Fan Y, Li W, Zhao X, Qi J, Huang H, Zhou D, Ning Z, Lu X. Results from a multicenter, open-label, pivotal phase II study of chidamide in relapsed or refractory peripheral T-cell lymphoma. Ann Oncol. 2015 Aug;26(8):1766-71. doi: 10.1093/annonc/mdv237. Epub 2015 Jun 23. PMID 26105599
- [Background] Zhang Q, Wang T, Geng C, Zhang Y, Zhang J, Ning Z, Jiang Z. Exploratory clinical study of chidamide, an oral subtype-selective histone deacetylase inhibitor, in combination with exemestane in hormone receptor-positive advanced breast cancer. Chin J Cancer Res. 2018 Dec;30(6):605-612. doi: 10.21147/j.issn.1000-9604.2018.06.05. PMID 30700929
- [Background] Jiang Z, Li W, Hu X, Zhang Q, Sun T, Cui S, Wang S, Ouyang Q, Yin Y, Geng C, Tong Z, Cheng Y, Pan Y, Sun Y, Wang H, Ouyang T, Gu K, Feng J, Wang X, Wang S, Liu T, Gao J, Cristofanilli M, Ning Z, Lu X. Tucidinostat plus exemestane for postmenopausal patients with advanced, hormone receptor-positive breast cancer (ACE): a randomised, double-blind, placebo-controlled, phase 3 trial. Lancet Oncol. 2019 Jun;20(6):806-815. doi: 10.1016/S1470-2045(19)30164-0. Epub 2019 Apr 27. PMID 31036468
- [Background] Sabnis GJ, Goloubeva OG, Kazi AA, Shah P, Brodie AH. HDAC inhibitor entinostat restores responsiveness of letrozole-resistant MCF-7Ca xenografts to aromatase inhibitors through modulation of Her-2. Mol Cancer Ther. 2013 Dec;12(12):2804-16. doi: 10.1158/1535-7163.MCT-13-0345. Epub 2013 Oct 3. PMID 24092810